CLINICAL TRIAL: NCT01508949
Title: NNC 90-1170 Mechanism of Action: A Single-centre, Randomised, Double-blind, Parallel-group, Placebo-controlled Trial Evaluating the Effect of NNC 90-1170 on Weight and Appetite in Obese Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide on Weight and Appetite in Obese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1333
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Once daily dosing of 0.6 mg for 8 weeks, injected subcutaneously
  Other Names: NNC 90-1170
  Arms: NNC 90-1170
Drug: placebo — Once daily dosing of 0.6 mg for 8 weeks, injected subcutaneously
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the effect of NNC 90-1170 (liraglutide) on weight and appetite in obese subjects with type 2 diabetes treated with diet and/or sulphonylurea or repaglinide.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Diet treated and/or subjects in monotherapy with sulphonylurea or repaglinide
* HbA1c for diet treated subjects 6.5-12%, both inclusive
* HbA1c for sulphonylurea or repaglinide treated subjects maximum 10%
* Body mass index (BMI) at least 27 kg/m^2
* Euthyroid subjects
* Fasting blood glucose 7-14 mmol/l

Exclusion Criteria:

* Impaired liver function
* Impaired renal function
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Recurrent severe hypoglycaemia as judged by the Investigator
* Known or suspected allergy to trial product or related products
* Use of any drug (except for OHAs (oral hypoglycaemic agents), which in the Investigator's opinion could interfere with the glucose level or body weight. Stable doses, for 3 months or greater, of thyroid hormone replacement are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-06; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Change in weight

SECONDARY OUTCOMES:
Total fat mass (assessed by use of DEXA (dual energy X-ray absorptiometry) scan)
Waist circumference
Spontaneous energy intake assessed in connection to the ad libitum lunch meal
Appetite assessed in connection with the fixed breakfast meal (assessed by the use of VAS (visual analogue scale))
Gastric emptying rate
Energy expenditure
HbA1c (Glycosylated Haemoglobin)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Frederiksberg C, Denmark

REFERENCES:
- [Result] Harder H, Nielsen L, Tu DT, Astrup A. The effect of liraglutide, a long-acting glucagon-like peptide 1 derivative, on glycemic control, body composition, and 24-h energy expenditure in patients with type 2 diabetes. Diabetes Care. 2004 Aug;27(8):1915-21. doi: 10.2337/diacare.27.8.1915. PMID 15277417
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com